CLINICAL TRIAL: NCT05386095
Title: The Motor Effect of 0.25%Bupivacaine Ultrasound Guided Axillary Block Versus 0.19% Bupivacaine Ultrasound Guided Axillary Block in Pediatrics Undergoing Below Elbow Orthopedic Surgeries: A Randomized Controlled Trial
Brief Title: Axillary Brachial Plexus Block Using 0.25% Bupivacaine Versus Using 0.19%Bupivacaine in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd elmoneim Adel Abd elmoneim, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-621-2021
Record Dates: First submitted 2022-05-13; First posted 2022-05-23 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Acute Postoperative Pain; Motor Activity
Keywords: postoperative pain; axillary brachial plexus block; below elbow orthopedic surgeries; Bupivacaine; motor sparing block
MeSH Terms: conditions — Pain, Postoperative; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.25%Bupivacaine group (Active Comparator): Axillary brachial plexus block will be done with patient in supine position under general anesthesia . A total volume of (0.5ml/kg) 0.25% bupivacaine + 1 µg/kg dexmedetomidine.this volume will be divided equally among the median,ulnar,radial and the musculocutaneous nerve.
  The surgical procedure will be start after 15-20 min. At the end of surgery, residual neuromuscular block will be antagonized with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg. All patients will receive 15mg/kg paracetamol IV.
  At recovery room motor power will be assisted using Modified Bromage scale , then each 30 min till full recover of motor power. post operative pain assessment will be done using (FLACC score) for Pain assessment.For patients with pain score more than 4\10 ,Pethidine I.V will be given as rescue analgesic (1 mg/kg) when needed and total rescue analgesia will be recorded.
  Interventions: Procedure: 0.25%Bupivacaine Axillary brachial plexus block
- 0.19%Bupivacaine group (Experimental): Axillary brachial plexus block will be performed with the patient in supine position under general anesthesia .
  A total volume of (0.5ml/kg) 0.19% bupivacaine + 1 µg/kg dexmedetomidine will be divided equally among the median,ulnar,radial and the musculocutaneous nerve.
  The surgical procedure will be start after 15-20 min.At the end of surgery, residual neuromuscular block will be antagonized with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg. All patients will receive 15mg/kg paracetamol IV.
  At recovery room motor power will be assessed using Modified Bromage scale , then each 30 min till full recover of motor power. post operative pain assessment will be done using (FLACC score) for Pain assessment,For patients with pain score more than 4\10 ,Pethidine I.V will be given as rescue analgesic (1 mg/kg) when needed and total rescue analgesia will be recorded..
  Interventions: Procedure: 0.19% Bupivacaine Axillary brachial plexus block

INTERVENTIONS:
Procedure: 0.25%Bupivacaine Axillary brachial plexus block — Axillary brachial plexus block will be induced with patient in supine position under GA with the linear probe ultrasound , the operating arm will be abducted by 70 , externally rotated, and the elbow will be flexed to ~90. Within the axillary crease the probe will be placed in sagittal position bounded by the pectoralis major antero-medially and the latissimus dorsi and teres major posteromedial. The median nerve lies between 9 and 12 o'clock position above the axillary artery and below the biceps muscle; (ii) the ulnar nerve located superficially between the axillary vein and artery (iii) the radial nerve lies above the conjoint tendon of the teres major and latissimus dorsi (iiii) The musculocutaneous nerve lies between biceps and coracobrachialis muscle .The block will be applied by 22 gag needles at cephalic side of the probe. A total volume of (0.5ml/kg) of 0.25% Bupivacaine plus 1 µg/kg dexmedetomidine will be used.this volume will be divided equally among the four nerves.
  Arms: 0.25%Bupivacaine group
Procedure: 0.19% Bupivacaine Axillary brachial plexus block — Axillary brachial plexus block will be induced with patient in supine position under GA with linear probe ultrasound , the operating arm will be abducted by 70 , externally rotated, and the elbow will be flexed to ~90. Within the axillary crease the probe will be placed in sagittal position bounded by the pectoralis major antero-medially and the latissimus dorsi and teres major posteromedial. The median nerve lies between 9 and 12 o'clock position above the axillary artery and below the biceps muscle; (ii) the ulnar nerve located superficially between the axillary vein and artery (iii) the radial nerve lies above the conjoint tendon of the teres major and latissimus dorsi (iiii) The musculocutaneous nerve lies between biceps and coracobrachialis muscle.The block will be applied by 22 gag needles at cephalic side of the probe. A total volume of (0.5ml/kg) of 0.19% Bupivacaine plus 1 µg/kg dexmedetomidine will be used.this volume will be divided equally among the four nerves.
  Arms: 0.19%Bupivacaine group

SUMMARY:
Postoperative pain is a common manifestation in orthopedic patients, mainly due to intraoperative tissue damage and inadequate intraoperative pain assessment and management .Axillary brachial plexus block provides motor and sensory block with the distribution of the median, radial, ulnar and musculocutaneous branches so can be conducted with upper limb orthopedic surgery in hand, rest and elbow surgery distal to the cubital fossa . In this study the investigators will investigate (0.19%) and (0.25%) bupivacaine for postoperative motor power recovery and post-operative analgesic efficacy in ultrasound guided axillary brachial plexus block among pediatric patient undergoing below elbow orthopedic surgery.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be randomly assigned to receive either:

(Group A: n=30)will receive 0.25% bupivacaine plus 1 µg/kg dexmedetomidine . (Group B: n=30) will receive 0.19% bupivacaine plus 1 µg/kg dexmedetomidine. Using computer generated number and concealed using sequentially numbered, sealed opaque envelope technique. There will be no restrictions or stratiﬁcations in the randomization process. The allocation envelope will be opened by the assistant lecturer at the time of anesthetic preparation.

All children will be anaesthetized in accordance with the local policy of the Abu El-Reesh pediatric hospital-Cairo university's pediatric anaesthetic unit. Except for oral clear liquids intake 2 hours before surgery, all children will fast for 6 hours. Patients will attend in the preparation room one hour before the operation to get a preoperative checkup, as well as their age and body weight will be recorded. Premedicated by intramuscular injection of atropine 0.02 mg/Kg and midazolam 0.2 mg/Kg . On arriving the operating room, heart rate (HR) ,oxygen saturation and non-invasive blood pressure will be continuously recorded, using standard monitor (Dräger infinity vista XL).

All patients will be induced with inhalational anesthetic using (100%) O2 + Sevoflurane. After deepening of the anesthesia, I.V. line will be inserted and atracurium 0.5mg/kg and fentanyl 1μg/kg patients will be given, then the patients will be intubated by appropriate size of endotracheal tube volume control ventilation (VCV) 5-7 ml/kg and respiratory rate will be adjusted to keep and PaCO2 levels between 30-35 mmHg using (G.E-Datex-Ohmeda, Avance CS2, USA) anesthesia machine. Anesthesia will be maintained with an isoflurane 1 MAC with 50% oxygen in air, with the goal of keeping the bispectral index (BIS) measurement between (40-60), and atracurium top-ups of 0.1mg/kg will be given every 30 minutes for neuromuscular blockade.

Axillary brachial plexus block will be conducted with the patient in supine position under general anesthesia.

In Group A:(0.25 %bupivacaine group) ultrasound guided Axillary brachial plexus block will be conducted using a total volume of 0.5ml/kg of bupivacaine 0.25% + 1 µg/kg dexmedetomidine.

In Group B:(0.19%bupivacaine group)ultrasound guided Axillary brachial plexus block will be conducted using a total volume of 0.5ml/kg of bupivacaine 0.19% + 1 µg/kg dexmedetomidine.

The surgical procedure will be start after 15-20 min. If there is an increase in heart rate or mean arterial blood pressure of more than 20% of the baseline value after skin incision then it will be considered as block failure and these patients will be excluded from the study. 1-2ug/kg intravenous fentanyl will be given to failed block.

At the end of surgery, residual neuromuscular block will be antagonized with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg. All patients will receive 15mg/kg paracetamol IV.

At recovery room motor power will be assisted using Modified Bromage scale by attending anesthesiologists who will be blinded to the study groups, then each 30 min till full recover of motor power .

The post operative pain assessment in the PACU and the ward, patient will be assessed immediately postoperatively and then at 1st, 4th, 8th, 12th hour post-operatively using (FLACC score) for Pain assessment.

ELIGIBILITY:
Inclusion Criteria:

1. American society of Anesthesiologists (ASA )class I-II
2. Duration of surgery less than 1 hour.

Exclusion Criteria:

1. Parent refusal.
2. Prolonged procedure exceeding 1 hour.
3. Patients with apparent infection at site of needle insertion.
4. Patients with any coagulation disorder(Platelets ≤ 50,000 and/or international normalized ratio INR> 1.5)
5. Patients with known neuropathy or brachial plexus injury.
6. Patients with any cardiac, hepatic, renal failure.
7. Patient with known sensitivity to local anesthetic drugs.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Motor power using modified bromage scale on admission to the PACU (post anesthesia care unit) | on admission to the PACU (10 minutes after extubation)
  Modified Bromage scale is a scale designed to assess degree of motor power as shown; Grade Definition 4 Full muscle strength in relevant muscle groups 3 Reduced strength, but able to move against resistance 2 Ability to move against gravity, but not against resistance
  1 Discrete movements (trembling) of muscle groups 0 Lack of movement

SECONDARY OUTCOMES:
Pain score at 0,1,2, 4, 8 and 12 hours postoperative. | 12 hours
  FLACC is a behavioral pain assessment scale used for nonverbal or preverbal patients who are unable to self-report their level of pain. Pain is assessed through observation of 5 categories including face, legs, activity, cry, and consolability.
cumulative 24 hours opioid consumption | 24 hours
  amount of pethidine given to the patient post operative(mg/24 hour)
intraoperative heart rate | every 15 minutes intraoperative till end of surgery (up to 1 hours)
  Heart rate of the patient intraoperatively (beat/minute)
intraoperative mean blood pressure | every 15 minutes intraoperatively till end of surgery (up to 1 hour)
  mean arterial blood pressure of the patient intraoperatively (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Maha G Hanna, professor, Principal Investigator — Anesthesia department , cairo university; Dalia S Abdelkader, assprofessor, Principal Investigator — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy Hospitals, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No